CLINICAL TRIAL: NCT01799109
Title: Lung Function Changes of Mild to Moderate Asthmatic Children Treated by Nebulized MgSO4
Brief Title: Lung Function of Asthmatic Children by Nebulized MgSO4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dai Jihong, professor, Chongqing Medical University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-2012CQ
Record Dates: First submitted 2012-11-23; First posted 2013-02-26 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Asthma
Keywords: magnesium sulfate; nebulization; lung function
MeSH Terms: conditions — Asthma | interventions — Magnesium Sulfate; Albuterol; Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- nebulization ms and albuterol (Experimental): magnesium sulfate 150mg & albuterol 2.5mg nebulized with 5-6L/min of oxygen and consisted about 5 min,which used only once
  Interventions: Drug: Magnesium Sulfate & albuterol
- nebulized albuterol (Active Comparator): albuterol 2.5mg nebulized with 5-6L/min of oxygen and consisted about 5 min,which used only once
  Interventions: Drug: albuterol
- nebulized ms (Experimental): magnesium sulfate 150mg nebulized with 5-6L/min of oxygen and consisted about 5 min,which used only once
  Interventions: Drug: magnesium

INTERVENTIONS:
Drug: Magnesium Sulfate & albuterol
  Arms: nebulization ms and albuterol
Drug: albuterol
  Arms: nebulized albuterol
Drug: magnesium
  Arms: nebulized ms

SUMMARY:
Asthma is a common chronic respiratory illness which results in frequent wheezing, cough,reduced quality of life. Standard treatment for asthma attack includes oxygen therapy, β2-agonists (e.g. albuterol) and inhaled anticholinergics and corticosteroids. Although inhaled short-acting β2-agonists (SAB) is the initial choice to control acute asthma exacerbation, there are still some asthmatic children unresponsive to this management. The Global Initiative in National Asthma (GINA) does not recommend intravenous magnesium sulfate (MgSO4) for routine use in asthma exacerbation especially in young children. But intravenous MgSO4 can reduce hospital admission rates in certain patients due to several effects e.g relaxation of smooth muscle,blocking acetylcholine. In addition,adding MgSO4 to nebulized SAB provides greater benefit in severe asthma exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* asthmatic children with controlled clinical manifestation

Exclusion Criteria:

* fever
* history of chronic disease like bronchopulmonary dysplasia or cystic fibrosis
* allergic to acetylcholine, albuterol or magnesium
* use any bronchodilator agents before the Clinic day

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
changes of lung function | 10minutes and 20minutes post-dose
  to observe changes of Forced expiratory volume in one second and peak expiratory flow in controlled asthmatic children after respectively nebulized MgSO4、albuterol and combination of MgSO4 and albuterol in lung function test.

SECONDARY OUTCOMES:
Nebulized magnesium sulfate alone effectively improve lung function | 10minutes and 20minutes post-dose
  After Ach challenge,FEV1 and PEF decreased in all three groups.But only in albuterol and magnesium group,they presented statistically significant while not in combination therapy group.After each intervention, FEV1 and PEF increased.But there was only statistically significant in FEV1 of magnesium and PEF of albuterol at 10 minutes and these two treatment at 20 minutes
the number of participants with adverse events as a measure of safety and tolerability | 20minutes
  to observe if anyone appear side effects such as nausea, vomiting, hypotension et al in patients who participating in our experiment. we did not found adverse reaction or other side effect in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Dai, professor, Study Director — Chongqing Medical University
Locations (1):
- Center of Respiratory Disorders,Children's Hospital,Chongqing medical university, Chongqing, Chongqing Municipality, China